CLINICAL TRIAL: NCT01591512
Title: A Prospective Longitudinal Collection of Subjects Diagnosed With Small Cell
Brief Title: A Prospective Longitudinal Collection of Subjects Diagnosed With Small Cell Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Decision was made by Sponsor to stop the trial.
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Collaborators: Medical Research Networx LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: FDI-36
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; SCLC; Lung Cancer; Subjects diagnosed with SCLC who will undergo treatment
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of whole blood and urine.

SUMMARY:
The purpose of this study is to collect samples to evaluate the ProGRP and NSE assays independently as aids for monitoring the course of disease and therapy in subjects diagnosed with SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Confirmed diagnosis of SCLC or mixed SCLC/non-SCLC per histopathology results
* Scheduled to undergo first-, second- or third-line treatment for SCLC, including chemotherapy, chemotherapy + radiation therapy, or combined concurrent chemoradiotherapy.
* Able to understand and willing to provide Informed Consent

Exclusion Criteria:

* No diagnosis of SCLC
* Not scheduled to undergo treatment for the diagnosis of SCLC
* Unable to provide Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Small cell lung cancer patients undergoing treatment.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Kelly Family Medical Center, PC, Eastpointe, Michigan
  - St.Louis Cancer Care, LLP, Bridgeton, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Hematology Oncology Consultants, Inc., St Louis, Missouri